CLINICAL TRIAL: NCT01960491
Title: Prospective Single Center Pilot Clinical Study to Evaluate the Safety and Effectiveness of an Intracardiac Septal Closure Device With Biodegradable Framework in Patients With Clinically Significant Atrial Septum Defect (ASD) or Patent Foramen Ovale (PFO)
Brief Title: FIH Study With CBSO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carag AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013.4678
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Atrial Septal Defect (ASD); Patent Foramen Ovale (PFO)
MeSH Terms: conditions — Heart Septal Defects, Atrial; Foramen Ovale, Patent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device Closure of Atrial Septal Defect (Experimental)
  Interventions: Device: Device Closure of Atrial Septal Defect

INTERVENTIONS:
Device: Device Closure of Atrial Septal Defect — Device Closure of Atrial Septal Defect by "Carag Bioresorbable Septal Occluder"

SUMMARY:
The objective of this study is to evaluate the effectiveness and the safety of the intracardiac septal closure device (CBO), as well as the practicability of implantation of this device using the accessories (DS for CBO).

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years - no upper limit of age
* Body weight > 40 kg
* Patients with an isolated ASD or PFO determined as suitable for closure via a commercially available device
* In ASD patients, echocardiographic evidence of right ventricular overload, and a stretched diameter of the defect up to 25 mm
* In patients with PFO, echocardiographic evidence of right to left shunt, and intraatrial tunnel length up to 4 mm
* Signed informed consent, respectively ability to give written informed consent after being told of the potential benefits and risks of entering the trial
* For female patients of child bearing capacity: Exclusion of pregnancy before start of the study and willingness to use adequate contraceptive methods to prevent pregnancy during the study

Exclusion Criteria:

* ASD/PFO larger than a stretched diameter of 25 mm, or defects unsuitable for percutaneous closure
* Intraatrial tunnel longer than 4 mm
* Multiple or fenestrated ASD, ostium primum or sinus venosus atrial septal defect, coronary sinus defect
* Any significant cardiac valve dysfunction
* Anomalous pulmonary veins
* Defects with inadequate margins, as is consistent with current standards of care, such that the device will not position appropriately so as to avoid interference with other cardiac structure, or that will subject the device to increased risk of embolization post deployment.
* Acquired pathological or congenital deficiencies of the cardiovascular system (any other than ASD; e.g. transposition of vessels, calcification, myocardial infarction, intracardiac thrombi), being clinically significant, respectively interfering in the investigator's opinion with the conduct of study
* Clinically significant dilated cardiomyopathy (paroxysmal or caused by e.g. myocarditis or other reasons)
* Any patient known to have extensive or complex congenital cardiac anomaly which can only be adequately repaired by way of cardiac surgery
* Echocardiographic evidence of thrombus in the left atrium, left atrial appendage, or other cardiac chamber, and in the inferior vena cava.
* Patients who within one month prior to implantation are known to have sepsis or any systemic infection that has not been successfully treated prior to device placement
* Active endocarditis or other infections producing bacteremia.
* Clinically relevant arrhythmia
* Patients whose vasculature, through which access to the defect is gained, is inadequate to accommodate the size of the device, the position controls or the introduction sheath
* Documented history of bleeding, clotting or coagulation disorders, untreated ulcer or any other contraindications to acetylsalicylic acid therapy, unless another anti-platelet agent can be administered for 6 months
* Known hypercoagulable state
* Anamnesis respectively diagnosis of pregnancy, or breastfeeding patients
* Any disorder in the investigator's opinion that could interfere with compliance or safety evaluation as well as any severe concurrent illness that would limit life expectancy (e.g. malignancies)
* Participation in an investigational drug or device trial within 30 days prior to selection (day 0) or current inclusion in any other clinical trial or research project
* Subjects who, in the opinion of the investigator, will be inappropriate for inclusion into this clinical trial or will not comply with requirements of the study
* Patients who are kept lawfully in an institution
* Clinical investigations shall be conducted in vulnerable populations only when they cannot be carried out in non-vulnerable populations and shall follow the additional ethics committee procedures where applicable. These clinical investigations shall be designed specifically to address health problems that occur in the vulnerable population, and offer the possibility of direct health-related benefit to the vulnerable population

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-05; Primary Completion 2017-01 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Effective closure of defect | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Horst Sievert, Prof. Dr., Principal Investigator — CardioVaskuläres Centrum Frankfurt, Germany
Locations (1):
- CardioVaskuläres Centrum, Frankfurt, Germany